CLINICAL TRIAL: NCT02176330
Title: Assessing the Impact of Using ePAQ on Quality and Cost of Patient Care in Uro-gynaecology: a Randomised Controlled Trial
Brief Title: Does Using a 'Virtual Clinic' in Urogynaecology Improve Patient Experience and Reduce Cost?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Georgina Jones, Reader in Social Science, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STH14733; North Sheffield Ethics 07/H130 (Other Grant/Funding Number: Sheffield Hospitals Charitable Trust 115512)
Record Dates: First submitted 2014-06-23; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pelvic Floor Disorders
Keywords: Randomised Controlled Trial; Virtual Clinic; ePAQ-PF; Pelvic Floor Disorders; Economic Analysis
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): ePAQ-PF followed by a face to face consultation.
  Interventions: Other: ePAQ-PF followed by a face to face consultation
- Virtual Clinic (Experimental): ePAQ-PF followed by a telephone consultation.
  Interventions: Other: ePAQ-PF followed by a telephone consultation.

INTERVENTIONS:
Other: ePAQ-PF followed by a telephone consultation. — All women randomised to this arm of the study were entered onto the hospital electronic patient record system under the ePAQ clinic. They were were posted an information letter and an epaq-online voucher inviting them to complete the questionnaire on-line. The clinician used these results along with the patient's own casenotes and original referral letter to support the subsequent consultation. The research nurse (HJW) then arranged their telephone consultation. Women in this group who felt unable to complete the questionnaire online would use this telephone call with the research nurse to make arrangements to attend and complete the questionnaire at the hospital.
  Arms: Virtual Clinic
Other: ePAQ-PF followed by a face to face consultation — All women randomised to this arm of the study were posted an appointment to attend the urogynaecology clinic. They were were posted an information letter and an epaq-online voucher inviting them to complete the questionnaire on-line. The clinician used these results along with the patient's own casenotes and original referral letter to support the subsequent consultation. Women then attended for their face to face clinic consultation as normal. Women in this group who felt unable to complete the questionnaire online were given the opportunity to complete the questionnaire at the hospital when they attended for their consultation.
  Arms: Usual care

SUMMARY:
The purpose of this study is to assess the impact of using a virtual clinic which combines a web-based interactive questionnaire (ePAQ-PF) used in advance of clinic appointments in combination with a telephone consultation has on patient experience and cost compared to standard care.

DETAILED DESCRIPTION:
ePAQ is a web-based interactive questionnaire (electronic pelvic floor assessment questionnaire) that provides a detailed evaluation of a woman's pelvic floor symptoms and their impact on her quality of life. Touch-screen technology has been combined with computer programming (Dot Net & SQL Server) and existing paper-based instruments to produce an interactive user-friendly system that facilitates immediate data entry, analysis and storage. The instrument has evolved during several years' collaborative work with colleagues in a range of disciplines, including Gynaecology, Medical Physics, Colorectal Surgery, Urology and General Practice, as well as involving a women's health user-group and regular surveys of patients' views.1 Research in primary and secondary care has established the psychometric properties of the instrument.2 The system has won a National award for innovation (HITEA) and was cited in Lord Warner's Annual Report on NHS Innovation.3 EPAQ Systems Ltd is one of the first NHS spin-out technology companies to be established in the UK (created jointly with Sheffield Teaching Hospitals NHS Trust in November 2006).

More recent development work has resulted in the creation of a website, where subjects can securely and anonymously access and use the ePAQ system via the Internet. This potentially allows subjects to use system in advance of clinic appointments (as opposed to the current practice of their completing it on arrival in clinic, immediately prior to their appointment). This study aims to evaluate the impact that using ePAQ in this way may have on the efficiency and quality of patient care. Initial survey data suggest that many women attending urogynaecology clinics do have access to the Internet and would be willing to use the system on-line & in advance of clinic appointments.4 The facility is also available in the Gynaecology Unit for women without Internet access to attend specifically for supervised use of the system. The in-depth assessment provided by the ePAQ may then be used to support an initial telephone consultation with a clinician, following which patients may be directed to the most appropriate clinic, as well as being provided with information and advice and have some forms of treatment initiated (such as behavioural therapy). The proposed randomised study aims to compare outcomes in women who use the ePAQ system in this way with women who undergo standard care in the Urogynaecology Unit.

The major advantage of electronic systems, when compared with paper questionnaires, relate to the practicalities of clinical data capture. Electronic questionnaires are comparable in terms of reliability and can be superior in terms of efficiency and response rate. In addition, electronic touch-screen questionnaires have been shown to be acceptable to patients, regardless of their age or educational background. Data quality is high, even in disadvantaged and technophobic subjects and cost analysis has shown potential economic advantages.5,6,7,8,9 Pelvic floor disorders in women, such as incontinence and prolapse, share common aetiologies and commonly coexist. Estimates vary, though it is estimated that approximately 20% of adult women experience regular urinary incontinence, 5% have some incontinence of faeces and 11% suffer with prolapse.10,11,12 However, despite better understanding of these conditions, bowel, bladder, vaginal and sexual dysfunction remain understandably taboo subjects and many women still regard them as inevitable consequences of childbirth and ageing. The personal cost to individuals is high, however simple and effective treatments are increasingly available. Many disorders respond well to behavioural, physical or medical therapy and such conservative treatments are generally recommended prior to consideration of invasive investigations or surgery.13 In clinical practice, clinical assessment is central to diagnosis and management and the restoration of function, with a view to improving quality of life, is the principal aim of treatment. It is well recognised that clinical interview data may be unreliable, being based on clinicians' rather than patients' views of their condition. It seems appropriate therefore, to seek ways of improving clinical assessment in order to enhance the quality of care and reliably measure outcome. Many women with pelvic floor disorders are managed in the community by GPs, nurses, physiotherapists or continence nurse advisors. In secondary and tertiary care, urologists, gynaecologists, colorectal surgeons and geriatricians are likely to be involved. However, at all levels, inconsistencies in clinical assessments represent an impediment to effective communication and the multidisciplinary approach advocated by the DoH, who in 2000 recommended the following:

* Full assessment leading to first line treatment in the primary care setting, with treatment & management plans agreed with individual patients.
* The provision of an integrated continence service, bringing together agreed protocols and procedures for primary, secondary and tertiary care.
* A comprehensive continence service, at home and in homes, bringing together all relevant health disciplines.

The further development of ePAQ has the potential to substantially augment this process by using on-line assessments to support patients' initial management and triage. Using ePAQ in advance of clinic appointments may provide patients and clinicians with prompt and valuable information and assist in directing patients to the most appropriate clinics in primary and secondary care. However, such a development warrants scrutiny in terms of patient experience and cost.

The ePAQ is now an established part of standard care and is in routine use in the Sheffield Urogynaecology Unit. All new patients are given the opportunity to complete the questionnaire, online, at home and their printed results are then used to inform the subsequent clinical consultation. The aims of this research are to measure the impact that using a virtual clinic (ePAQ-PF in advance of clinic appointments + a telephone consultation) has on patient care and cost compared to standard care (ePAQ-PF in advance of clinic appointments + a face to face consultation).

ELIGIBILITY:
Inclusion Criteria:

* All women referred to Sheffield Teaching Hospitals urogynaecology services, aged > 18 and able to read and understand English will be eligible to enter the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The Patient Experience Questionnaire | This was posted to patients at one time point. This was posted no longer than two weeks after patients had attended for their first clinic consultation (Baseline).
  The primary outcome measure was the Patient Experience Questionnaire (PEQ) [1] completed after the patients first clinical consultation. The PEQ was developed and validated specifically to measure patients' experience of interaction, emotion and consultation outcome. It contains 16 items in four dimensions, including 1) communication, 2) emotions, 3) short-term outcome, and 4) barriers. Three of the scales are scored from 1-5, and the emotions scales runs from 1 to 7. A high score represents a good communication experience, positive emotions, positive consultation outcome and a lack of communication barriers.

SECONDARY OUTCOMES:
The Client Satisfaction Questionnaire-8. | This was posted to patients at one time point. This was posted no longer than two weeks after patients had attended for their first clinic consultation (Baseline).
  A modified version of the CSQ-8 was administered (Howie et al, 1997; 1998). This validated instrument contains 8 items measuring the patient's satisfaction following a consultation asking 1) how they rate the service, 2) did they get the service they wanted, 3) to what extent the service me their needs, 4) would they recommend the service to their friends, 5) how satisfied they were with the amount of help received, 6) if the services received helped then to deal more effectively with their problems, 7) overall satisfaction with the service and 8) if they would return to the services if they required help again. The CSQ-8 is a eight-item self-complete questionnaire, which generates a score with a 8 to 32 range, with a higher score indicating more patient satisfaction.
The Short-Form-12 | A subset of patients were asked to complete the SF-12 at two time points. This was posted after their intervention i.e. first consultation (Baseline) and six months later (Time 2).
  The SF-12 is a standardised, multidimensional, generic measure of health related quality of life (HRQOL), and was administered to patients at baseline and 6 months post initial consultation. The results from the SF-12 can be converted into utilities using the SF-6D (Brazier & Roberts 2004). These are a value anchored on a scale of 0 (death) to 1 (full health) which represent individuals preference for a health condition. These values are assigned to health states and combined with the number of years spent in that health state to calculate quality adjusted life years (QALY) which are needed for cost utility analyses.
The QQ-10 | This was posted to patients at one time point. This was posted no longer than two weeks after patients had attended for their first clinic consultation (Baseline).
  The QQ-10 is a 10-item instrument specifically designed for evaluating patients views on the value and burden of using of a questionnaire as part of their healthcare (Moores et al, 2012)
The Number and Type of Referrals | Data collected at the six month follow-up (Time 2)
  The total number and individual type of referrals made were used to evaluate the impact of ePAQ on the referral patterns and clinical visits made within the continence care pathway. At 6-month follow-up we will measure the number and type of referrals made on behalf of that patient; i.e. primary care (community nursing, community physiotherapy, GP, district nurse, practice nurse) and secondary care (gynaecology, urology, colorectal surgery, physiotherapy). These data will be collected in both groups using a standard proforma.

OTHER OUTCOMES:
Resource Use Proforma | Data collected at the six month follow-up (Time 2).
  The primary economic analysis will estimate the NHS costs of providing assessment and care up to six months in both arms of the study, and cost effectiveness by an incremental cost per quality-adjusted life year (QALY). These costs will include the costs of using ePAQ + telephone consultations, referrals, prescriptions (drugs / appliances / pads) and treatments. A broader societal costing will also be undertaken to consider costs to the patients and the economy in terms of private expenditure and time taken off work, respectively. These additional data will be in the standard proforma posted to both groups of patients at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina L Jones, D.Phil, Principal Investigator — University of Sheffield
Locations (1):
- The Jessop Wing Hospital, Sheffield, South Yorkshire, United Kingdom